CLINICAL TRIAL: NCT00017186
Title: Phase II Study of Gemcitabine and Epirubicin for the Treatment of Mesothelioma
Brief Title: Gemcitabine and Epirubicin in Treating Patients With Malignant Mesothelioma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCTG-N0021; NCCTG-N0021; CDR0000068659 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 2001-06-06; First posted 2003-01-27 (Estimated); Last update posted 2016-12-07 (Estimated); Status verified 2016-12

CONDITIONS: Malignant Mesothelioma
Keywords: localized malignant mesothelioma; advanced malignant mesothelioma; recurrent malignant mesothelioma
MeSH Terms: conditions — Mesothelioma, Malignant | interventions — Epirubicin; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- gemcitabine + epirubicin (Experimental): Patients receive gemcitabine IV over 30 minutes on days 1 and 8 and epirubicin IV on day 1. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients achieving complete response (CR) receive 2 additional courses beyond CR.
  Quality of life is assessed at baseline, prior to course 3, at 3 months, and then at 1 year.
  Patients are followed every 3 months for 1 year, every 4 months for 1 year, and then every 6 months for 3 years.
  Interventions: Drug: epirubicin hydrochloride; Drug: gemcitabine hydrochloride

INTERVENTIONS:
Drug: epirubicin hydrochloride
Drug: gemcitabine hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combining gemcitabine and epirubicin in treating patients who have malignant mesothelioma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the antitumor activity of gemcitabine and epirubicin in patients with malignant pleural mesothelioma.
* Determine the toxicity of this regimen in this patient population.
* Determine the time to progression and overall survival of patients treated with this regimen.
* Assess quality of life in patients treated with this regimen.

OUTLINE: This is a multicenter study.

Patients receive gemcitabine IV over 30 minutes on days 1 and 8 and epirubicin IV on day 1. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients achieving complete response (CR) receive 2 additional courses beyond CR.

Quality of life is assessed at baseline, prior to course 3, at 3 months, and then at 1 year.

Patients are followed every 3 months for 1 year, every 4 months for 1 year, and then every 6 months for 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed malignant pleural mesothelioma
* At least 1 measurable lesion that can be accurately measured in at least one dimension

  * At least 20 mm (2 cm) in diameter

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* At least 12 weeks

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* AST no greater than 3 times ULN

Renal:

* Creatinine no greater than 1.5 times ULN

Cardiovascular:

* LVEF at least 50%
* No history of congestive heart failure
* No New York Heart Association class III or IV heart disease

Other:

* No uncontrolled infection
* No other severe underlying disease that would preclude study participation
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer, noninvasive carcinomas, or localized prostate cancer
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 6 months after study participation

PRIOR CONCURRENT THERAPY:

Chemotherapy:

* No more than 1 prior chemotherapy regimen for malignant pleural mesothelioma
* No prior gemcitabine or anthracyclines

Other:

* No concurrent cimetidine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2001-07; Primary Completion 2004-08 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
time to progression | Up to 5 years

SECONDARY OUTCOMES:
survival | Up to 5 years
quality of life | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Scott Okuno, MD, Study Chair — Mayo Clinic
Locations (24):
- United States (24):
  - MBCCOP - Gulf Coast, Mobile, Alabama
  - CCOP - Mayo Clinic Scottsdale Oncology Program, Scottsdale, Arizona
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - CCOP - Cedar Rapids Oncology Project, Cedar Rapids, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - Siouxland Hematology-Oncology, Sioux City, Iowa
  - CCOP - Wichita, Wichita, Kansas
  - CCOP - Ochsner, New Orleans, Louisiana
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - CCOP - Duluth, Duluth, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Coborn Cancer Center, Saint Cloud, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Medcenter One Health System, Bismarck, North Dakota
  - CCOP - Merit Care Hospital, Fargo, North Dakota
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - CCOP - Geisinger Clinic and Medical Center, Danville, Pennsylvania
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - CCOP - Sioux Community Cancer Consortium, Sioux Falls, South Dakota
  - CCOP - St. Vincent Hospital Cancer Center, Green Bay, Green Bay, Wisconsin

REFERENCES:
- [Background] Huschka MM, Mandrekar SJ, Schaefer PL, Jett JR, Sloan JA. A pooled analysis of quality of life measures and adverse events data in north central cancer treatment group lung cancer clinical trials. Cancer. 2007 Feb 15;109(4):787-95. doi: 10.1002/cncr.22444. PMID 17211864
- [Result] Okuno SH, Delaune R, Sloan JA, Foster NR, Maurer MJ, Aubry MC, Rowland KM Jr, Soori GS, Nikcevich DA, Kardinal CG, Northfelt DW, Adjei AA; North Central Cancer Treatment Group. A phase 2 study of gemcitabine and epirubicin for the treatment of pleural mesothelioma: a North Central Cancer Treatment Study, N0021. Cancer. 2008 Apr 15;112(8):1772-9. doi: 10.1002/cncr.23313. PMID 18224661